CLINICAL TRIAL: NCT05474729
Title: The Efficacy and Safety of Minocycline for Chronic Autoimmune Uveitis
Brief Title: Minocycline for Chronic Autoimmune Uveitis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dan Liang, Dan Liang, PhD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MINOCU
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Minocycline; Uveitis; Retinal Degeneration
MeSH Terms: conditions — cyclopia sequence; Uveitis; Retinal Degeneration | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: minocycline capsule
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- minocycline (Experimental): minocycline capsule 100mg per day orally
  Interventions: Drug: minocycline

INTERVENTIONS:
Drug: minocycline — minocycline capsule 100mg per day orally

SUMMARY:
Autoimmune uveitis is one kind of non-infectious, sight-threatening, relapsing and severe ocular disease. Approximately 20%-25% autoimmune uveitis patients suffer from the dilemma of blindness for the chronic and persistent inflammatory state in the eyes, which results in continuous destroy in the structure of the eyes and gradually leads to irreversible damage on visual function. However, it shows limiting efficacy of current treatment including glucocorticoids, immunosuppressant and biologics for chronic autoimmune uveitis. Minocycline has been regarded to have anti-apoptosis and immunemodulatory function for decades and it has been illustrated to be beneficial in several neuro-degenerative and neuro-inflammatory diseases. This trial aims to investigate the efficacy and safety of minocycline for chronic autoimmune uveitis with retinal degenerative changes.

ELIGIBILITY:
Inclusion Criteria:

* Participant diagnosed of autoimmune diseases with visual function damage (decrease of BCVA, loss of retinal structure)
* Participant aged from 18-60 years old.
* Participant that signed the informed consent document and is able to complete the following visits.

Exclusion Criteria:

* Participant is allergy to minocycline or tetracyclines.
* Participant has no contraindications of minocycline or tetracyclines.
* Participant has an abnormal function of liver, heart, kidney and thyroid.
* Participant is using glucocorticoids, immunosuppressants or biologics.
* Female that is pregnant, breast-feeding or planning to become pregnant.
* Participant that is currently using other medications for other diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of macular sensitivity | At 6 and 12 months
  Change of macular sensitivity measured by MAIA
Change of BCVA | At 6 and 12 months
  Change of BCVA measured by ETDRS
Change of Visual field | At 6 and 12 months
  Change of Visual field measured by HVF 30-2 visual field testing
Changes in Implicit Time and Amplitude of Photopic and Scotopic Responses | At 6 and 12 months
  Changes in Implicit Time and Amplitude of Photopic and Scotopic Responses measured by Electroretinogram (ERG) Testing

SECONDARY OUTCOMES:
Change of macular vessel | At 6 and 12 months
  Change of macular vessel measured by OCTA
Change of Contrast Sensitivity | At 6 and 12 months
  Change of Contrast Sensitivity measured by F.A.C.T
Change of Color Visual | At 6 and 12 months
  Change of Color Visual measured by FM100
Change of QoL questionaire | At 6 and 12 months
  Change of QoL measured by VFI-25
Number of ocular and non-ocular adverse events Number of ocular and non-ocular adverse events Number of ocular and non-ocular adverse events Number of ocular and non-ocular adverse events Number of Ocular and Non-ocular Adverse Events | At 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dan Liang, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided